CLINICAL TRIAL: NCT06547047
Title: Effects of Speed, Agility, and Quickness Training on Physical, Cognitive, and Skill Performance Among University Soccer Major Students in China
Brief Title: Speed, Agility, and Quickness Training
Acronym: SAQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SUN MIN (Other)
Responsible Party: Sponsor-Investigator, SUN MIN, PhD Candidates, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMin
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Speed; Agility; Quickness; Physical Performance
Keywords: physical fitness; cognitive abilities; soccer skills; Sports performance
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: This study employs a parallel design in which participants are randomly assigned to two independent groups: the intervention group and the control group. Throughout the study, participants in the intervention group will undergo a 12-week Speed, Agility, and Quickness (SAQ) training program, conducted three times a week, each session lasting 60 minutes, including 15-20 minutes for warm-up and cool-down. Participants in the control group will continue with their regular training regimen. Tests will be conducted before, during, and after the intervention to assess changes in physical, cognitive, and skill performance. This parallel design ensures a clear evaluation of the SAQ training effects and minimizes confounding variables due to differences in training time and content.
Who Masked: Outcomes Assessor
Masking Description: In this study, both the participants and the outcomes assessor will be blinded to the group assignments to prevent bias. Participants will not be informed whether they are receiving SAQ training or regular training, and the outcomes assessor will also be unaware of the group assignments to ensure objective evaluation of the results. Care providers and investigators involved in administering the training sessions will know the group assignments due to the nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: SAQ Training (Experimental): Participants in the experimental group will undergo Speed, Agility, and Quickness (SAQ) training three times per week, with each session lasting 60 minutes, for a duration of 12 weeks. The training intensity will range from 70% to 100% of the participants' maximum effort. This program is designed to enhance physical fitness, cognitive abilities, and soccer-specific skills.
  Interventions: Behavioral: Speed, Agility, and Quickness (SAQ) Training
- Control Group: Regular Training (Active Comparator): Participants in the control group will engage in their regular training routine, which does not include the specific SAQ training regimen. The training intensity for the control group will also range from 70% to 100% of the participants' maximum effort. This routine will last for 12 weeks, with training sessions occurring three times per week for 60 minutes each session.
  Interventions: Behavioral: Regular Training

INTERVENTIONS:
Behavioral: Speed, Agility, and Quickness (SAQ) Training — The SAQ training will include exercises designed to improve speed, agility, and quickness, such as ladder drills, cone drills, sprint drills, and reaction drills.
  Arms: Experimental Group: SAQ Training
Behavioral: Regular Training — Participants in the control group will follow a standard soccer training regimen, which includes general conditioning exercises, skill drills, and tactical training.
  Arms: Control Group: Regular Training

SUMMARY:
This study aims to evaluate the effects of Speed, Agility, and Quickness (SAQ) training on the physical, cognitive, and skill performance of university soccer major students in China. The hypothesis is that SAQ training will significantly improve students' physical fitness (e.g., speed, agility), cognitive functions (e.g., reaction time, decision-making), and soccer skills (e.g., ball control, passing). The study will recruit 52 university soccer major students, randomly assigned to an intervention group and a control group, with 26 students in each group. The study will last for 12 weeks, and tests will be conducted before, during, and after the intervention. The expected outcome is that the intervention group will show superior performance in various tests compared to the control group, thereby validating the effectiveness of SAQ training.

DETAILED DESCRIPTION:
This study adopts a cluster randomized controlled trial (CRCT) design to evaluate the impact of SAQ training on the physical, cognitive, and skill performance of university soccer major students. The study will recruit 52 eligible university soccer major students, randomly assigned to the intervention group and the control group, with 26 students in each group. The study will last for 12 weeks, with the intervention group undergoing SAQ training three times a week, while the control group continues their regular training.

The SAQ training program includes the following components:

Warm-up and Cool-down: Each training session begins and ends with a 10-minute warm-up and cool-down to ensure safety.

Training Content: The SAQ training includes speed runs, agility exercises, and quick reaction drills, each session lasting 60 minutes.

Assessment Metrics: The study will assess students' physical fitness (speed, agility), cognitive functions (reaction time, decision-making), and soccer skills (ball control, passing).

Testing Time Points:

Pre-test: Initial assessment of all participants before the intervention. Mid-test: Mid-term assessment after 6 weeks of intervention. Post-test: Final assessment after the completion of the intervention.

Data Collection and Analysis:

Data Collection: Standardized testing methods will be used to assess all participants before, during, and after the intervention.

Data Analysis: Data will be analyzed using SPSS software, employing independent sample t-tests and ANOVA to compare differences between the intervention and control groups across various metrics.

Quality Assurance and Data Validation:

Quality Assurance Plan: An independent quality control team will oversee data collection and entry to ensure accuracy and completeness.

Data Validation: Data will be validated by comparing it with external sources (e.g., medical records, paper reports) to ensure authenticity and representativeness.

Sample Size Estimation and Statistical Analysis Plan:

Sample Size Estimation: Based on preliminary studies, the required sample size is estimated to be 52 to ensure statistical significance of the results.

Statistical Analysis Plan: Multivariate regression analysis and other methods will be used to control for confounding variables and analyze the impact of SAQ training on various metrics in detail.

ELIGIBILITY:
Inclusion Criteria

* Male soccer major students (age ≥18 years old)
* At least 3 years of professional soccer training
* No recent history of surgery or injury
* No participation in SAQ training programs within 8 weeks prior to the study
* Able to provide written informed consent and willing to participate in the entire study and complete all assessments

Exclusion Criteria

* Recent history of fractures or other injuries
* Currently participating in an SAQ training program

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Flexibility | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by the sit-and-reach test. Results are recorded in centimeters (cm), with higher scores indicating better flexibility.
Agility | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by the Arrowhead Agility Test. Results are recorded in seconds (s), with shorter times indicating better agility.
Sprint | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by sprints at 5m, 10m, 20m, and 30m. Results are recorded in seconds (s), with shorter times indicating better speed.
Upper Body Strength | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by pull-ups. Results are recorded as the number of completed pull-ups, with more pull-ups indicating greater upper body strength.
Lower Limb Explosiveness | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by vertical jump. Results are recorded in centimeters (cm), with higher jump heights indicating greater explosiveness.
Aerobic Endurance | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by the Yo-Yo Intermittent Recovery Test Level 2 (Yo-Yo2). Results are recorded as maximum distance covered（m）, with higher distances indicating better aerobic endurance.
Reaction Time | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by a computerized reaction time test. Results are recorded in milliseconds (ms), with shorter reaction times indicating faster responses.
Selective attention | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Through the computer flanker task, the results are recorded in milliseconds (ms), with higher accuracy and shorter reaction time indicating better decision-making ability.
Dribbling Agility | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  Measured by the 22-meter slalom dribble test. Results are recorded in seconds (s), with shorter times indicating better dribbling skills.
Passing performance | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  When measuring passing performance using the Loughborough Soccer Passing Test (LSPT), results are recorded as total time and passing accuracy. Total time is measured in seconds (s) and includes the time from the start of the test to the completion of the last pass, including all penalty time. Shorter total times indicate better performance. Passing accuracy is recorded by the number of successful passes into target areas, with more successful passes indicating better passing skills. Penalties are applied as follows: five seconds for completely missing the target area or passing to the wrong target, three seconds for missing the target area, three seconds for handling the ball, two seconds for passing from outside the designated area, and two seconds for the ball touching any cone.

SECONDARY OUTCOMES:
Height | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  The height of the participant is recorded, typically measured to two decimal places, in meters (m).
Weight | Pre-intervention: Week 0 Mid-intervention: Week 6 Post-intervention: Week 12
  The weight of the participant is recorded, measured to one decimal place, in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Min Sun, Principal Investigator — FACULTY OF EDUCATIONAL STUDIES
Locations (1):
- Faculty of Educational Studies, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared. The data is intended solely for research purposes and will only be accessible to the research team. Data confidentiality will be maintained, and no individual data will be made available to external parties.

REFERENCES:
- [Background] Brown, L., & Ferrigno, V. (2014). Training for speed, agility, and quickness, 3E. Human Kinetics
- [Background] Lee YS, Lee D, Ahn NY. SAQ training on sprint, change-of-direction speed, and agility in U-20 female football players. PLoS One. 2024 Mar 13;19(3):e0299204. doi: 10.1371/journal.pone.0299204. eCollection 2024. PMID 38478514
- [Background] Trecroci A, Cavaggioni L, Rossi A, Moriondo A, Merati G, Nobari H, Ardigo LP, Formenti D. Effects of speed, agility and quickness training programme on cognitive and physical performance in preadolescent soccer players. PLoS One. 2022 Dec 1;17(12):e0277683. doi: 10.1371/journal.pone.0277683. eCollection 2022. PMID 36454889
- [Background] Treisman, A. (1977). Focused attention in the perception and retrieval of multidimensional stimuli. Perception & psychophysics, 22, 1-11
- [Background] Development of speed, agility, and quickness for the female soccer athlete.
- [Background] Zamanzadeh V, Ghahramanian A, Rassouli M, Abbaszadeh A, Alavi-Majd H, Nikanfar AR. Design and Implementation Content Validity Study: Development of an instrument for measuring Patient-Centered Communication. J Caring Sci. 2015 Jun 1;4(2):165-78. doi: 10.15171/jcs.2015.017. eCollection 2015 Jun. PMID 26161370
- [Background] Milanovic Z, Sporis G, Trajkovic N, James N, Samija K. Effects of a 12 Week SAQ Training Programme on Agility with and without the Ball among Young Soccer Players. J Sports Sci Med. 2013 Mar 1;12(1):97-103. eCollection 2013. PMID 24149731
- See also: The physical fitness measurement indicators of this study refer to the Chinese Football Association's release of the "Stage Evaluation Standards for the Athletic Ability of Chinese Male Youth Players (2021 Edition)" — https://www.thecfa.cn/qttz/20220222/30316.html